CLINICAL TRIAL: NCT03686605
Title: The Edmonton Symptom Assessment System (ESAS) as a Screening Tool for Depression in Cancer Pain Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suratsawadee Wangnamthip, Lecturer, Mahidol University
Other Study IDs: Si 276/2018
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Screening Tool for Depresion in Cancer Pain Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer pain patients
  Interventions: Other: Thai version of the Edmontom Symptom Assessment System (ESAS)

INTERVENTIONS:
Other: Thai version of the Edmontom Symptom Assessment System (ESAS) — Screening and diagnostic questionaire for depression
  Other Names: Thai version of the Hospital Anxiety and Depression Scale (HADS); Thai version of 2Q; Thai version of the Mini International Neuropsychiatric Interview (M.I.N.I.); Thai version of the Diagnostic and Statistical Manual (DSM-5)

SUMMARY:
Compare Thai versions of the Edmonton Symptom Assessment System (ESAS) and the Hospiral Anxiety and Depression Scale (HADS) with Diagnostic and Statistical Manual (DSM-5), as a screening tool for depression in cancer pain patients

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who follow up as out patient at pain clinic, Siriraj hospital
* Age older than 18 years old
* Fluently read, write and speak in Thai language
* No cognitive impairment

Exclusion Criteria:

* Unstable clinical presentation
* Severe pain or pain numerical rating scale more than 7
* Severe associated symptoms such as nausea, vomiting
* The patient who do not know their diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer pain patients
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Reliability and validity of Thai version of ESAS | 1 year
  Cut-off point, sensitivity, specificity, positive predictive value and negative predictive value of Thai version of ESAS

SECONDARY OUTCOMES:
Correlation of Thai version of ESAS, HADS and DSM-5 | 1 year
  Pearson correlation, Sperman rank correlation
Internal consistency of Thai version of ESAS and HADS | 1 year
  Cronbach's alpha

CONTACTS AND LOCATIONS:
Overall Officials: Suratsawadee Wangnamthip, MD, Principal Investigator — Lecturer
Locations (1):
- Faculty of medicine Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No